CLINICAL TRIAL: NCT03511872
Title: Peers Versus Professional Training of Basic Life Support in Syria: a Randomized Controlled Trial
Brief Title: Peers Vs Professionals in Basic Life Support Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2210110616
Record Dates: First submitted 2018-04-12; First posted 2018-04-30 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Basic Life Support Training Course
Keywords: Basic life support; cardiopulmonary resuscitation; medical undergraduate students; crisis; randomized controlled trial.

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with blinded assessors on medical students from the pre-clinical years (1st to 3rd years in Syria) at Syrian Private University. Students are randomly assigned to peer-led or to professional-led training group for one-day-course of basic life support skills.
Who Masked: Outcomes Assessor
Masking Description: Two blinded 10-year experienced professionals in emergency training (trainers in the Syrian resuscitation council) are asked to evaluate students' skills independently A third assessor who is also professional in emergency training is asked to resolve conflict judgments between live and camera assessment when existed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peers' group (Experimental): 36 Medical students are allocated randomly to Peers' group where they are trained on BLS skills by senior students.
  Four students from the latest three years of study in medical schools in Syria (4th, 5th, and 6th) are randomly selected and enrolled to be instructors for basic life support training course to transfer the resuscitation skills to medical students from pre-clinical years.
  Interventions: Other: Basic life support training
- Professionals' group (Experimental): 36 students are allocated randomly to professionals' group where they are trained on BLS skills by professional trainers in emergency. Four professionals (2 emergency doctors, cardiologist and anesthesiologist) are leading training to the control group to deliver the basic life support training course with the same duration and content as the intervention group.
  Interventions: Other: Basic life support training

INTERVENTIONS:
Other: Basic life support training — A course design was made to be consistent with ERC guidelines with local modifications made by emergency professionals in duration, instructor-to-trainee ratio, course materials, methods to deliver these materials theoretically, and the type of the manikin used to practice CPR. One-day-course consisting of 75, 20, 20, 20 minutes for theoretical BLS, chocking, recovery position, the practical representation of BLS scenario respectively followed by 40-minute practical training on BLS skills for each subgroup. Both arms of the study follow the same timeline and no extra time is given to any group.
  Same manikins were used for the training and the assessment. On the day of the experiment students in each arm are divided into 4 subgroups of maximum 9 students, each led by two trainers of BLS skills with a maximum ratio of 2 instructors to 9 students per group.

SUMMARY:
An Evaluation of Peer-led basic life support training course compared with professional-led course in a limited resource environment; A randomized controlled trial

DETAILED DESCRIPTION:
Peer training has been identified as a useful tool for delivering undergraduate training in basic life support (BLS) which is fundamental as an initial response in cases of emergency.

This study aimed to (1) Evaluate the efficacy of peer-led model in basic life support training among medical students in their first three years of study, compared to professional-led training and (2) To assess the efficacy of the course program and students' satisfaction of peer-led training.

A randomized controlled trial with blinded assessors will be conducted on 72 medical students from the pre-clinical years (1st to 3rd years in Syria) at Syrian Private University. Students will be randomly assigned to peer-led or to professional-led training group for one-day-course of basic life support skills.

Analysis will be done on students who underwent checklist based assessment using objective structured clinical examination design (OSCE) (practical assessment of BLS skills) and answered BLS knowledge checkpoint-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Medical student from 1st, 2nd and third year at Syrian Private University.
* Sign the consent form.

Exclusion Criteria:

* presence of any health problems preventing students from doing physical exercise.
* any serious acute or chronic illness (infectious, psychological, physical).
* scheduling conflict between the date of the BLS course and other faculty's classes or exams.
* missing the course or the assessment for any reason.
* refusing to sign the consent and having any prior experience in BLS skills (previously trained on BLS).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
BLS practical skills | Training and assessment were held at the same day of the experiment for both groups, 1) within 24 hours of providing the bls training course.
  A practical simulated scenario assessment using a checklist based evaluation in objective structured clinical examination (OSCE) design. The checklist is constructed in accordance to European resuscitation council (ERC) guideline. Students should perform each point correctly to pass the assessment (1- Safe approach, 2- call for help, 3- opening airway, 4-checking cardiopulmonary situation, 5- call ambulance, 6- CPR with effective depth, 7-rate and 8-position, 9-rescue breaths).

SECONDARY OUTCOMES:
BLS knowledge questionnaire | Training and assessment were held at the same day of the experiment for both groups. 1) within 24 hours of providing the bls training course.
  a 20-item questionnaire with 3 checkpoints per item (60-point-scale) derived from ERC materials after testing the applicability of the questionnaire by a pilot study.
Students' evaluation of BLS course survey | Training and assessment were held at the same day of the experiment for both groups. 1) within 24 hours of providing the bls training course.
  Students' reported outcomes using American Heart Association (AHA) survey of BLS course evaluation. This survey aims to investigate students' satisfaction and their opinions about the course.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Association AH. ECC Course Evaluation. 2012.
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Charlier N, Van Der Stock L, Iserbyt P. Peer-assisted Learning in Cardiopulmonary Resuscitation: The Jigsaw Model. J Emerg Med. 2016 Jan;50(1):67-73. doi: 10.1016/j.jemermed.2015.04.002. Epub 2015 Jun 20. PMID 26099910
- [Background] Fujiwara T, Nishimura M, Honda R, Nishiyama T, Nomoto M, Kobayashi N, Ikeda M. Comparison of peer-led versus professional-led training in basic life support for medical students. Adv Med Educ Pract. 2011 Jul 26;2:187-91. doi: 10.2147/AMEP.S22948. Print 2011. PMID 23745089
- [Background] Perkins GD, Hulme J, Bion JF. Peer-led resuscitation training for healthcare students: a randomised controlled study. Intensive Care Med. 2002 Jun;28(6):698-700. doi: 10.1007/s00134-002-1291-9. Epub 2002 Apr 24. PMID 12107673